CLINICAL TRIAL: NCT05288231
Title: Cardiac Manifestation in Adolescent After Pfizer COVID-19 Injection in Thailand
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chayasin Mansanguan, Associate Professor, Mahidol University
Other Study IDs: Cardiac and pfiizer
Record Dates: First submitted 2022-03-17; First posted 2022-03-21 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Covid-19 Vaccine
Keywords: pfizer-BioNTech Covid-19 vaccine; adult; Thailand; myocarditis; cardiac manifestation; Covid-19 vaccine
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic of ECG — All participants who enrolled in the study will be performed ECG, cardiac enzyme and echocardiography
  Other Names: Diagnostic of cardiac enzyme; Diagnostic of echocardiography

SUMMARY:
Rationale Recently, a CDC advisory Committee on Immunization Practices identified a likely association between the 2 COVID-19 mRNA vaccines from Pfizer-BioNTech and Moderna and cases of myocarditis and pericarditis. For the cardiovascular system, 4863 adverse events (AEs) were reported from the Pfizer vaccine. Common findings observed with vaccines under study were tachycardia(16.41%), flushing (12.17%), hypertension (5.82%), hypotension (3.6%), and increased heart rate (9.03%). In this study we characterized, classified, evaluate the dynamic of cardiac function and ECG abnormality after the Pfizer vaccine injection.

This is a prospective cohort study. All participants aged 13-18 years old and above who visited the second dose Pfizer covid-19 vaccine injection to determine cardiac manifestation.

Methods for analyzing research data The data will be collected from students enrollment at Kong thabbok upatham changkol kho so tho bo school and Wachirathamsatit school. The participant's history, physical exam, and laboratory data will be reviewed and data will be extracted based on the case record form (CRF). All data will be stored securely and analyzed using the SPSS® Statistics Version 23 developed by IBM®. Data entry will be carried out using coding and verification. Quantitative data will be expressed as mean with standard deviation (SD) or median (IQR) and qualitative data will be presented as a number of observations with percentage (%). Descriptive statistics will be used to summarize the baseline values and demographic data.

All p-values will be derived using the 2-tailed testing, and statistical significance will be set at 0.05 probability. All the categorical variables will be analyzed using the chi-square (x2) or Fisher's exact test whichever is appropriate. Normality of the distribution will be tested for the continuous variable using the Kolmogorov- Smirnov test. All the variables with normal distributions will be compared using the independent t-test and will be reported as mean ± standard deviation (SD). The variables that do not pass the normality test will be compared by means of the Mann-Whitney U test and will be reported as the median and interquartile range (IQR).

DETAILED DESCRIPTION:
Data Collection Methods

1. Participants' demographics will be collected at baseline using case record form.
2. Laboratory tests include: at 3 clinical visits (Baseline, Day3, Day7 and Day 14 (optional if have cardiac manifestation) after 2nd dose of Pfizer COVID-19 vaccine) 2.1. Cardiac biomarker (Troponin-T, CK-MB) 2.2. Echocardiography 2.3. ECG (Electrocardiography)

After getting approval from the Ethics Committee and before the start of the trial, the study team informed the interesting participants about the study by invitation letter with ZOOM or line meeting. Informed consent printed to the parents who interested in this project and bring to the team investigator before enrollment. A contact address and phone number will be provided for the interesting participants to call for more information about the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-18 years old
2. Both males and females
3. Received 1st dose Pfizer COVID-19 vaccine injection

Exclusion Criteria:

1. Unable to obtain written informed consent from the participants or their legal representatives
2. History of cardiomyopathy, tuberculous pericarditis, and constrictive pericarditis
3. Severe allergic reaction to COVID-19 vaccine

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Student age 13-18 who received 1st dose of pfizer COVID-19 vaccine from
  1. Kong thabbok upatham changkol kho so tho bo school
  2. Wachirathamsatit school
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participant with cardiac manifestation after Pfizer COVID-19 vaccine injection at baseline | Day 0
  cardiac manifestation defined as sinus tachycardia, hypertension at baseline
Number and percentage of participant with cardiac manifestation after Pfizer COVID-19 vaccine injection at day 3 | Day 3
  cardiac manifestation defined as sinus tachycardia, hypertension at day 3
Number and percentage of participant with cardiac manifestation after Pfizer COVID-19 vaccine injection at day 7 | Day 7
  cardiac manifestation defined as sinus tachycardia, hypertension at day 7

SECONDARY OUTCOMES:
Number and percentage of participant with Myocarditis after Pfizer COVID-19 vaccine injection at baseline | Day 0
  frequency (%) of participant with myocarditis at baseline
Number and percentage of participant with Myocarditis after Pfizer COVID-19 vaccine injection at day 3 | Day 3
  frequency (%) of participant with myocarditis at day 3
Number and percentage of participant with Myocarditis after Pfizer COVID-19 vaccine injection at day 7 | Day 7
  frequency (%) of participant with myocarditis at day 7
Number and percentage of participant with pericarditis after Pfizer COVID-19 vaccine injection at baseline | Day 0
  frequency (%) of participant with pericarditis at baseline
Number and percentage of participant with pericarditis after Pfizer COVID-19 vaccine injection at day 3 | Day 3
  frequency (%) of participant with pericarditis at day 3
Number and percentage of participant with pericarditis after Pfizer COVID-19 vaccine injection at day 7 | Day 7
  frequency (%) of participant with pericarditis at day 7
Number and percentage of participant abnormal cardiac biomarker after Pfizer COVID-19 vaccine injection at baseline | Day 0
  frequency (%) of participant with abnormal cardiac biomarker (Troponin and CKMB) at baseline
Number and percentage of participant abnormal cardiac biomarker after Pfizer COVID-19 vaccine injection at day 3 | Day 3
  frequency (%) of participant with abnormal cardiac biomarker (Troponin and CKMB) at day 3
Number and percentage of participant abnormal cardiac biomarker after Pfizer COVID-19 vaccine injection at day 7 | Day 7
  frequency (%) of participant with abnormal cardiac biomarker (Troponin and CKMB) at day 7

CONTACTS AND LOCATIONS:
Overall Officials: Chayasin Mansanguan, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Tropical Medicine, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data or leftover specimens will be shared for future study ONLY subjects who consent allow using their specimens. Sharing will be done without specimen identification.
Supporting Information: Study Protocol, ICF
Time Frame: 2 years after publication

REFERENCES:
- [Derived] Mansanguan S, Charunwatthana P, Piyaphanee W, Dechkhajorn W, Poolcharoen A, Mansanguan C. Cardiovascular Manifestation of the BNT162b2 mRNA COVID-19 Vaccine in Adolescents. Trop Med Infect Dis. 2022 Aug 19;7(8):196. doi: 10.3390/tropicalmed7080196. PMID 36006288